CLINICAL TRIAL: NCT02743390
Title: Effects of the TNF-alpha Inhibiton on Blood Pressure, Hemodynamic Parameters and Biomarkers in Resistant Hypertension
Brief Title: Effects of the TNF-alpha Inhibiton on Hemodynamic Parameters in Resistant Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Heitor Moreno Junior, Principal investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2015171517
Record Dates: First submitted 2016-04-05; First posted 2016-04-19 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Hypertension
Keywords: blood pressure; inflammation; tumor Necrosis Factor-alpha
MeSH Terms: conditions — Hypertension; Inflammation | interventions — Infliximab; Tumor Necrosis Factors; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNF-alpha inhibitor drug (Active Comparator): Infliximab infusion (TNF-α inhibitor, 3 mg/kg, 250mL)
  Interventions: Biological: Infliximab
- Placebo drug (Placebo Comparator): Saline infusion (250mL)
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Infliximab — Monoclonal antibody biologic drug that inhibits tumour necrosis factor alpha (TNF-α), 3 mg/kg for 2 hours (250mL)
  Other Names: Tumour necrosis factor alpha (TNF-α) inhibitor
  Arms: TNF-alpha inhibitor drug
Other: Saline — Saline for 2 hours (250mL)
  Arms: Placebo drug

SUMMARY:
Resistant hypertension (RH) is characterized by high blood pressure (BP) in spite of concurrent use of three or more antihypertensive agents of different classes, combined at optimal doses. Currently it has been largely discussed the influence of inflammation in RH. The BP variation promotes increased expression of pro-inflammatory cytokines, such as tumor necrosis factor-alpha, interleukins 1 and 6. It was showed that treatment with TNF-α inhibitor improves BP and endothelial function, and reduces arterial stiffness in patients with rheumatoid arthritis. Recently, it was demonstrated that TNF-α levels are increased in RH subjects compared to normotensives. This study aims to assess whether the acute inhibition of TNF-α changes hemodynamic parameters, such as mean BP levels in RH.

DETAILED DESCRIPTION:
This crossover, double-blind study will include 12 resistant hypertensive subjects - regularly followed at the Outpatient Resistant Hypertension Clinic/UNICAMP - which will randomized assigned to (1) saline infusion followed by infliximab infusion (TNF-α inhibitor, 3 mg/kg) and (2) infliximab followed by saline, for two hours and washout of the 40-day period between both infusions. It is expected that the TNF-α inhibition regulates hemodynamic parameters, such as mean BP, cardiac Output, total peripheral resistance, which may allow a better rational approach for the RH treatment.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis recommended by the AHA Statment on Resistant Hypertension (2008)
* a 6-month period clinic follow-up
* give written informed consent form

Exclusion Criteria:

* secondary Hypertension
* pseudoresistance hypertension (poor medication adherence and white coat hypertension)
* patients with symptomatic ischemic heart disease, impaired renal function, liver disease and history of stroke, myocardial infarction and peripheral vascular diseases
* pregnant women
* smoking
* autoimmune diseases

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure in mmHg | 15 minutes
  Mean blood pressure will be simultaneously assessed for 15 minutes in baseline, during and post the infusions

SECONDARY OUTCOMES:
Cardiac hypertrophy in g/m² | Baseline and post-1 week of the infusions
  Left ventricular mass index will be determined by echocardiography in baseline and post-1 week of the infusions
Endothelial function in percentage | Baseline and post-1 week of the infusions
  Endothelial function will be assessed by flow-mediated dilation in baseline and post-1 week of the infusions
Arterial stiffness in m/s | Baseline and post-1 week of the infusions
  Arterial stiffness will be determined by pulse wave velocity in baseline and post-1 week of the infusions
Tumor necrosis factor-alpha in pg/mL | Baseline and post-1 week of the infusions
  Plasma concentration of tumor necrosis factor-alpha will be determined by ELISA
Interleukin-6 | Baseline and post-1 week of the infusions
  Plasma concentration of Interleukin-6 will be determined by ELISA
Interleukin-10 | Baseline and post-1 week of the infusions
  Plasma concentration of Interleukin-10 will be determined by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula Faria, PhD, Study Chair — University of Campinas
Locations (1):
- University of Campinas (UNICAMP), Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided